CLINICAL TRIAL: NCT02628041
Title: A Phase II Randomized Trial Evaluating Acute and Late Toxicity of High-Dose Rate Brachytherapy and Low-Dose Rate Brachytherapy as Monotherapy in Localized Prostate Cancer
Brief Title: HDR Brachytherapy vs. LDR Brachytherapy Monotherapy in Localized Prostate Cancer
Acronym: HDRvsLDR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Université de Montréal (Other); Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Lara Hathout, MD, FRCPC, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-20-2016-2570
Record Dates: First submitted 2015-12-07; First posted 2015-12-11 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Prostate Cancer
Keywords: High-Dose-Rate Brachytherapy; HDR Monotherapy; LDR monotherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Permanent Iodine-125 seed implant (Active Comparator): Prostate brachytherapy using Iodine-125 seed implant to a prescription dose of 144 Gy delivered to the Target volume defined as Clinical Target volume (CTV)+ 0-3 mm margin.
  Interventions: Radiation: Permanent Iodine-125 seed implant
- High-dose-Rate Prostate brachytherapy (Experimental): Prostate brachytherapy implant using Iridium-192 to a prescription dose of 19 Gy delivered to the CTV in one fraction. Greater than 95% coverage of the CTV with the prescription dose is considered per protocol, 90-95% coverage is considered a minor deviation and, < 90% coverage is considered a major deviation.
  Attempts should be made to achieve these other dosimetric values:
  * D90: 105-115%
  * V150 ≤ 35%
  * V200 ≤ 12%
  Interventions: Radiation: High-Dose-rate Prostate Brachytherapy

INTERVENTIONS:
Radiation: Permanent Iodine-125 seed implant — Permanent Iodine seed implant is performed under general or epidural anesthesia with the patient is positioned in the lithotomy position.
  A Foley catheter is inserted in the bladder. Under transrectal ultrasound guidance, the prostates is scanned and the dosimetry is generated. Catheters are inserted in the prostate and the seeds are injected using the Nucletron automatic after loader according to the dosimetry plan.
  The catheters are removed at the end of the procedure.
  Arms: Permanent Iodine-125 seed implant
Radiation: High-Dose-rate Prostate Brachytherapy — High-Dose-Rate Prostate brachytherapy is performed under general or epidural anesthesia, the patient is positioned in the lithotomy position.
  A Foley catheter is inserted in the bladder. Under transrectal ultrasound guidance, catheters are inserted in the prostate to assure adequate coverage. The patient is returned in dorsal decubitus and a CT scan or Ultrasound scan is performed. A inverse-planning dosimetry plan is generated to deliver 19 Gy to the target volume. The patient is treated and then the implant is removed and anesthesia is reversed.
  Other Names: HDR implant
  Arms: High-dose-Rate Prostate brachytherapy

SUMMARY:
High-dose rate brachytherapy (HDRB) used as monotherapy is emerging as an alternative to Low-Dose Rate brachytherapy (LDRB) with excellent PSA-progression free survival as high as 90-100% for favorable prostate cancer at a median follow-up of 3-5 years.

HDRB has many advantages over LDRB such as prospective dosimetry not impacted by setup errors, organ motion and prostate swelling during treatment delivery. In addition, HDRB causes less acute and late urinary toxicity compared with LDRB. Acute urinary retention can lead to prolonged catheterization, pericatheter urine leakage, urinary tract infection and Trans-Urethral Resection of the Prostate resulting in diminished quality of life (QOL) and increased psychological distress.

The goal of the investigators' phase II randomized study is to evaluate the differences in QOL in the urinary domain between patients with favourable intermediate risk or extensive low-risk prostate cancer treated with LDRB and HDRB at 3 months using the Expanded Prostate Cancer Index Composite (EPIC) QOL scores. The 3 months cut-off endpoint has been chosen since HDRB-induced urinary toxicity subsides at 12 weeks compared to 12 months with LDRB. Secondary objectives include: bowel and sexual domain EPIC scores and International Prostate Symptom Score. The absolute PSA nadir and a prostate biopsy at 36 months will be reported to assess local control.

DETAILED DESCRIPTION:
Primary Endpoint:

• To evaluate the differences in QOL in the urinary domain between patients treated with Low-Dose Rate Brachytherapy (LDRB) and High-Dose Rate Brachytherapy (HDRB) at 3 months.

Secondary Endpoints:

* To compare LDRB vs. HDR as related to the Expanded Prostate Cancer Index Composite (EPIC) score in the bowel and sexual domain at baseline, 1, 3, 6, 12, and 24 months.
* To evaluate differences in urinary function using the IPSS which, will be filled in by the patient at baseline, 1, 3, 6, 12 and 24 months after the procedure.
* To report acute and long-term urinary, sexual and gastro-intestinal toxicity using the Common Terminology Criteria for Adverse Events (CTCAE) version 4 at each patient's visit.
* To report the dose to the bladder neck defined as 5 mm around the Foley catheter from the bottom of the Foley balloon to the prostatic urethra with a volume of at least 2 cc.
* To assess local control by performing prostate rebiopsy after radiotherapy at 36 months to assess treatment outcome.
* The absolute Prostate Specific Antigen ( PSA) nadir value will be reported as a secondary objective by PSA measurements every 6 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

-Histologically confirmed adenocarcinoma of the prostate diagnosed within the last 9 months.

Patients on active surveillance with evidence of disease progression are eligible to the protocol as long as they meet the eligibility criteria and have a recent prostate biopsy (within 9 months).

* Low-risk disease defined as: Clinical stage T1-T2 and Gleason 6 and PSA≤20 ng/mL.
* Intermediate-risk disease defined as: Clinical stage T1-T2 and Gleason 7 (3+4) and PSA ≤ 20 ng/mL and ≤ 60% of positive cores.
* Lymph node evaluation by either CT or MRI is optional and is left at the discretion of the treating physician.
* No alpha reductase inhibitors use within 2 weeks of randomization. A washout period of 2 weeks is required prior to randomization.
* Eastern Cooperative Oncology Group status 0-1
* No hormonal therapy is accepted.
* Prostate volume by Trans-rectal Ultrasound (TRUS) ≤ 60 cc.
* Internation Prostate Symptom Score (IPSS) ≤ 20 (alpha blockers allowed)

Exclusion Criteria:

* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, or other solid tumours curatively treated with no evidence of disease for ≥ 5 years.
* Prior or current bleeding diathesis
* Previous androgen deprivation therapy within 6 months of the registration.
* Radical surgery for carcinoma of the prostate, prior pelvic radiation, prior chemotherapy for prostate cancer, prior Transurethral resection of the prostate (TURP), prior cryosurgery of the prostate.
* Evidence of metastatic disease (radiology investigations at the discretion of the treating physician).
* Any serious active or co-morbid medical conditions, laboratory abnormality, psychiatric illness, active or uncontrolled infections, or serious illnesses or medical conditions that would prevent the patient from participating or to be managed according to the protocol (according to investigator's decision).
* Gleason score 7 (4+3), clinical stage≥ T3a, PSA > 20 and > 60% of positive cores.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-10; Primary Completion 2017-12 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Quality of Life differences at 3 months using the Expanded Prostate Cancer Index Composite in the urinary domain. | 3 months

SECONDARY OUTCOMES:
Quality of life differences using the Expanded Prostate Cancer Index Composite (EPIC) score in the bowel and sexual domain at baseline, 1, 3, 6, 12, and 24 months. | 24 months
Differences in urinary function using the International Prostate Symptom Score which, will be filled in by the patient at baseline, 1, 3, 6, 12 and 24 months after the procedure. | 24 months
Acute and long-term urinary, sexual and gastro-intestinal toxicity using the Common Terminology Criteria for Adverse Events (CTCAE) version 4 at each patient's visit. | 24 months
The dose to the bladder neck defined as 5 mm around the Foley catheter from the bottom of the Foley balloon to the prostatic urethra with a volume of at least 2 cc. | 1month
Local control by performing transrectal-ultrasound guided 12-core prostate rebiopsy at 36 months to assess treatment outcome. | 36 months
The absolute PSA nadir value will be reported as a secondary objective by PSA measurements every 6 months after the procedure. | every 6 months up to 5 years
  Patients will undergo a prostate biopsy at 36 months and the pathology will be reviewed by a Genito-urinary pathology expert and classified in 3 categories: negative (no evidence of cancer), positive ( persistence of cancer cells) and undetermined.

CONTACTS AND LOCATIONS:
Overall Officials: Lara Hathout, MD, FRCPC, Principal Investigator — Centre Hospitalier Universitaire du CHU de Québec
Locations (1):
- CHU de Québec- L'Hôtel-Dieu de Québec, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided